CLINICAL TRIAL: NCT04962009
Title: A 90-Day, Open-Label, Multi-Site, Pilot Study Evaluating the Safety and Intraocular Lowering Effect of Delivering Travoprost Using a Punctal Plug Delivery System (Evolute®) in Subjects With Elevated Intraocular Pressure
Brief Title: Safety and Intraocular Lowering Effect of Delivery of Travoprost Evolute® in Subjects With Elevated Intraocular Pressure
Status: Completed | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGLA-2021-01
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Elevated Intraocular Pressure (IOP)
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Travoprost Evolute (Travoprost Punctal Plug Delivery System), 166 ug
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug (Experimental): Each subject will have his/her lower puncta of each eye inserted with a Travoprost Evolute®. Each study subject will be instructed to return to the investigator's office the next day, 7, 28, 60 and 90-days after the insertion of their plugs for follow-up examinations.
  Interventions: Combination Product: Travoprost Evolute® (Travoprost Punctal Plug Delivery System), 166 ug

INTERVENTIONS:
Combination Product: Travoprost Evolute® (Travoprost Punctal Plug Delivery System), 166 ug — Each subject will have his/her lower puncta of each eye inserted with a Travoprost Evolute®. Each study subject will be instructed to return to the investigator's office the next day, 7, 28, 60 and 90-days after the insertion of their plugs for follow-up examinations.

SUMMARY:
This is a pilot, open-label, multi-center clinical study. Each potential subject that has met all screening inclusion/exclusion criteria will undergo a six-week washout phase where they will discontinue the use of their topical hypotensive medication.

After the six-week washout, each potential subject will return for a baseline visit. Investigators will verify that a potential subject has discontinued the use of their topical hypotensive medication(s) and all their prohibited systemic medications for the last 6 weeks. In addition, each subject will have discontinued the use of all other ocular drops, gels or ointments 24 hours prior to the visit (Visit 2) and continues to meet all screening and washout criteria. After completing the baseline examination, each potential subject that meet all baseline inclusion/exclusion for the treatment phase of the study will have his/her lower puncta of each eye inserted with a Travoprost Evolute®. Each study subject will be instructed to return to the investigator's office the next day, 7, 28, 60 and 90-days after the insertion of their plugs for follow-up examinations.

DETAILED DESCRIPTION:
This is a pilot, open-label, multi-center clinical study. Each potential subject that has given HIPAA and informed consent and has meet all screening inclusion/exclusion criteria will undergo a six-week washout phase where they will discontinue the use of their topical hypotensive medication. In addition, during the washout phase, each potential study subject will also discontinue the use of all prohibited systemic medications.

After the six-week washout, each potential subject will return for a baseline visit (Visit 2). Investigators will verify that a potential subject has discontinued the use of their topical hypotensive medication(s) and all their prohibited systemic medications for the last 6 weeks. In addition, each subject will have discontinued the use of all other ocular drops, gels or ointments 24 hours prior to the visit (Visit 2) and continues to meet all screening and washout criteria. After completing the baseline examination, each potential subject that meet all baseline inclusion/exclusion for the treatment phase of the study will have his/her lower puncta of each eye inserted with a Travoprost Punctal Plug Delivery System (Evolute®). Each study subject will be instructed to return to the investigator's office the next day, 7, 28, 60 and 90-days after the insertion of their plugs for follow-up examinations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, 18 years of age or older at the time of the screening examination and has been diagnosed with bilateral OAG or OH
2. A subject must be able and willing to read, comprehend and give authorization for Use/Disclosure of Health Information (HIPAA) and informed consent
3. A subject must not have taken any ocular hypertension medication(s) within the last 12 hours of the screening visit unless in the opinion of the screening physician it poses an undue risk.
4. A subject must be willing to have the lower puncta of each eye inserted with a study plug
5. A subject's screening visit (pre-washout) Intraocular Pressures (IOPs), measured between 8:00 and 10:00 AM, is less than 22 mmHg in both eyes
6. A subject Intraocular Pressures (IOPs) are currently controlled (< 22 mm Hg) with a topical prostaglandin or in conjunction with one other topical ocular hypotensive drug, not including any fixed-combination formulations (i.e., Cosopt, Combigan, Azarga, etc.), in both eyes for at least one month
7. A subject has a Best-Corrected Distance (Glasses), pinhole visual acuity of 20/100 (Snellen) or better in both eyes
8. A subject has documented perimetry results within the last 6 months prior to the Screening Visit for both eyes NOTE: If perimetry measurement are older than 6 months, perform automated perimetry at the screening visit

Exclusion Criteria:

1. A subject with a history of non-response to topical prostaglandin eye drops for OAG/OH
2. A subject with angle-closure glaucoma, neovascular glaucoma, traumatic glaucoma or iridocorneal endothelium syndrome in either eye
3. A subject with a known sensitivity to travoprost, fluorescein, topical anesthetic, silicone, any inactive ingredient of the Travoprost Evolute® or any other products required for study procedures
4. A subject with a history of complications, AEs, trauma or disease in the nasolacrimal area, whether or not it was due to punctal plug wear, including but not limited to dacryocystitis, inflammation or canaliculitis in either eye
5. A subject with a history of intolerance to punctal plugs or a known sensitivity to any inactive ingredient of the punctal plug, silicone, topical anesthetic, or any other products required for the study
6. A subject with structural lid abnormalities (i.e., ectropion, entropion) in either eye
7. A subject with an active lid disease in either eye (i.e., moderate or severe blepharitis, meibomianitis) that requires medical treatment
8. A subject with any clinically significant (moderate or severe) lid, conjunctival or corneal findings in either eye at the screening visit
9. A subject with a history of chronic/recurrent inflammatory eye disease (i.e., scleritis, uveitis, herpes keratitis) in either eye
10. A subject who would require the use of any ocular medication(s), an over-the-counter drop(s), ointment(s) or gel(s), other than the study hypotensive medication(s) in either eye during the study period
11. A subject who has had any ophthalmic surgical procedures (i.e., glaucoma laser, minimally invasive glaucoma surgery, cataract, refractive, etc.) in either eye within the last six months or will require ophthalmic surgery before completing the study
12. A subject with a history of penetrating keratoplasty in either eye
13. A subject requiring the use of a contact lens in either eye at any time during the study period
14. A subject with advanced diabetic retinopathy, branch retinal vein occlusion or central retinal vein occlusion in either eye
15. A subject with a history of macular edema in either eye
16. A subject currently on any systemic medication [i.e., beta-blocker, carbonic anhydrase inhibitors, corticosteroids (including dermal), etc.] that may have an effect on the subject's Intraocular Pressure (IOP), or who will require its use during the study period
17. A subject with an uncontrolled systemic disease or a medical condition that may increase the risk associated with study participation or administration of study treatment or that may interfere with the interpretation of study results (e.g., autoimmune disease if the subject is on chronic medications and has ocular involvement; host-versus-graft disease)
18. A subject currently participating or has participated within the last 30 days prior to the start of this study in a drug, device or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stiles Eyecare Excellence, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Intraocular Pressure (IOP) Change
Description: Mean percent change in Intraocular Pressure (IOP) from baseline to days 90
Time Frame: day 90
Measure: Mean (Full Range); unit: mean % Intraocular Pressure (IOP) change
Arm/Group | Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug
Number analyzed (Participants) | 10
mean % Intraocular Pressure (IOP) change | -14.6 [-36.1 to 7.6]

ADVERSE EVENTS:
Time Frame: AEs data was collected at all timepoints from baseline to 90 days (final visit)
Description: AEs were collected by the investigator asking the patient "Have you had any problems since your last visit?" and collecting the response
Arm/Group | Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travoprost Evolute® (Travoprost Punctal Plug Delivery System, T-PPDS), 166 ug (N=12)
Foreign Body sensation, single/mild (Eye disorders) | 1 (1)
retinal migraine OS (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can not publish data without our permission. Sponsor can change communication and extend an embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04962009/Prot_SAP_000.pdf